CLINICAL TRIAL: NCT05315063
Title: Comparison of Muscle Energy Technique and Eccentric Training on Hamstring Flexibility in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01208 Mehwish Iqbal
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: muscle energy technique; eccentric training; hamstring flexibility; active knee extension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric Training (Experimental): Once achieved, this flexed hip position will be held for 5 seconds. This procedure will be repeated 6 times with no rest between repetitions
  Interventions: Other: Eccentric Training; Other: Muscle Energy Technique (PIR)
- Muscle Energy Technique (PIR) (Experimental): muscle energy technique
  Interventions: Other: Eccentric Training; Other: Muscle Energy Technique (PIR)

INTERVENTIONS:
Other: Eccentric Training — Once achieved, this flexed hip position will be held for 5 seconds. This procedure will be repeated 6 times with no rest between repetitions
Other: Muscle Energy Technique (PIR) — The participant will be asked to resist the movement with no more than 25% of strength. The contraction will be held for 7-10 seconds followed by complete relaxation of the limb.
  On exhalation, the knee joint will be straightened (extended) towards its new barrier and through that barrier a stretch was applied and maintained for 30 seconds.3 repetitions of this process will be done

SUMMARY:
Flexibility is the ability of a muscle to lengthen and allow one joint (or more than one joint in series) to move through a full range of motion (ROM).Adequate flexibility is important to maintain balance, agility and musculoskeletal function. A decrease in muscular flexibility does not only reduces functional level of individual but also causes musculoskeletal injuries. Loss of muscle flexibility or muscle tightness is decreased ability of a muscle to lengthen which results in decreased ROM,and for hamstring reduced flexibility is the inability to achieve more than 160 degree of knee extension while the hip is flexed at 90 degree.

Muscle energy technique (MET) is an manual technique developed by osteopaths and is now used in many different manual therapy professions, to treat soft tissue, mobilize joints, stretch tight muscles and fascia, reduce pain and to improve circulation and lymphatic drainage.

Eccentric training allows the muscle to elongate naturally, this elongation is achieved by having the subjects eccentrically contract the antagonist muscle to move the joint through the full available range in slow controlled manner.

DETAILED DESCRIPTION:
Flexibility is the ability of a muscle to lengthen and allow one joint (or more than one joint in series) to move through a full range of motion (ROM). Adequate flexibility is important to maintain balance, agility and musculoskeletal function. A decrease in muscular flexibility does not only reduces functional level of individual but also causes musculoskeletal injuries. Loss of muscle flexibility or muscle tightness is decreased ability of a muscle to lengthen which results in decreased ROM. and for hamstring reduced flexibility is the inability to achieve more than 160 degree of knee extension while the hip is flexed at 90 degree. Hamstring muscles have a great tendency to shortening even in normal circumstances, due to their multi-joint function and their tonic postural character. Techniques previously investigated for hamstring flexibility include static, ballistic and active assisted stretching exercise, ice, heat, soft tissue massage, ultra sound, Short Wave Diathermy, myofascial release, (PNF), kinesio taping, MET Each of these interventions has demonstrated clinical and experimental success; no agreement has been reached on a standard protocol for treatment.

Muscle energy technique (MET) is an manual technique developed by osteopaths and is now used in many different manual therapy professions, to treat soft tissue, mobilize joints, stretch tight muscles and fascia, reduce pain and to improve circulation and lymphatic drainage.

Eccentric training allows the muscle to elongate naturally, this elongation is achieved by having the subjects eccentrically contract the antagonist muscle to move the joint through the full available range in slow controlled manner. Eccentric resistance exercise may prevent injury to the muscle tendon unit by improving the muscle's ability to absorb more energy before failing and it is a better training strategy to improve the flexibility as it also increases strength and protects against muscle damage.

ELIGIBILITY:
Inclusion Criteria:

• A deficit of >20° of knee extension with the hip at 90°

Exclusion Criteria:

* lower extremities pathology.
* any history of hamstring injuries.
* acute or chronic low back pain.
* history of lower limb fracture.
* surgery of hamstring or back.
* pelvis, hip or knee deformity.
* Involved in any stretching routine

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test | two weeks
  Active knee extension test is an objective test for measuring flexibility/tightness of hamstring muscles with goniometer. Every subject is set in recumbent position with hip and knee flexed in 90°.A wooden box is utilized to keep up the correct position of hip. The pelvis is strapped down to the table for stabilization and controlling any accessory movement and the participant's head is kept in a neutral position to avoid any neural tension. For goniometer the landmarks used are the greater trochanter of the femur, lateral femoral condyle and lateral malleolus. The subject is then asked to extend the dominant lower extremity as far as possible until a mild stretch sensation is felt and a full circle goniometer is then used to measure the angle. Assessment to be done at baseline,3rd session and 6th session.
Sit and Reach Test: | two weeks
  The test involves sitting on the floor with back and head against the wall, legs stretched out straight ahead. Shoes are removed and the sole of feet are placed flat against the box. Both knees should be locked and pressed flat on the floor with the palms facing downwards and the hands-on top of each other. Subject reaches forward along the measuring line as far as possible. assessment to be done at baseline,3rd session and 6th session.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Rawal Institute of Rehabilitation Sciences, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No